CLINICAL TRIAL: NCT03747263
Title: Individualized Approach vs. Fixed Approach Utilizing the Novel Arctic Front Advanced Pro Cryoballoon for Pulmonary Vein Isolation in Patients With Paroxysmal Atrial Fibrillation: A Randomized Observational Trial
Brief Title: Individualized Approach vs. Fixed Approach
Acronym: INDI-FREEZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Christian-H. Heeger, MD, Consultant Rhythmology, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-256
Record Dates: First submitted 2018-10-29; First posted 2018-11-20 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Freeze-Catheter ablation (Experimental): The individualized "time-to-effect" protocol utilizing the AFA-Pro applies a freeze-cycle until documentation of PVI based on continuous real-time recordings from the Achieve catheter inside the PV. After documentation of PVI the freeze-cycle is prolonged for additional 90 seconds. If no PVI is achieved after 90 seconds or a temperature of -<30° is not reached after 40 seconds the freeze cycle is stopped, the cryoballoon will be repositioned to possibly achieve a better position. Afterwards the freeze-cycle will be restarted. If no real-time PV signal recording can be obtained, a standard freeze-cycle of 180 seconds is applied. No bonus-freeze-cycle is applied in this protocol.
  Interventions: Procedure: Catheter ablation
- Fixed Freeze-Catheter ablation (Active Comparator): The fixed-freeze-cycle protocol utilizing the AFA-Pro comprises a fixed freeze-cycle duration of 180 seconds. If PVI is not achieved with the first freeze-cycle, another 180 seconds freeze-cycle will be applied until documented PVI. After PVI no bonus freeze-cycle is applied.
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Electrophysiology studies are performed during conscious sedation using boluses of midazolam and fentanyl and a continuous infusion of propofol. Vital parameters are continuously monitored. One 7F standard diagnostic catheter is positioned inside the coronary sinus (CS) via the femoral vein. One 8,5-F sheath is advanced to the left atrium (LA). After transseptal catheterization, intravenous heparin is administered to target an activated clotting time of ≥300 seconds. PV angiographies are obtained for each PV and PV recordings are registered at baseline in SR. The 8.5F transseptal sheath (TS) is changed over the wire for a 12F steerable TS.
  Other Names: Cryoballoon

SUMMARY:
The purpose of the current study is to assess differences regarding the acute efficacy, safety, procedural duration, radiation exposure and long-term success of the novel AFA-Pro in combination of an individualized shortened ablation protocol containing a reduced freezing time to the standard approach of a fixed ablation protocol in patients with symptomatic PAF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* The patient understands the nature of the study, treatment procedure and provides written informed consent
* Symptomatic paroxysmal atrial fibrillation as defined by the current guidelines
* Willing to comply with specified pre-, post- and follow-up testing, evaluations and requirements
* Expected to remain available (geographically stable) for at least 12 months after enrollment

Exclusion Criteria:

* Atrial fibrillation secondary to a reversible cause or of non-cardiac origin
* Previous AF ablation procedure
* Longstanding persistent AF
* Documented left atrial thrombus on imaging (e.g., transesophageal echocardiogram, angiogram)
* NYHA functional Class IV heart failure
* Unstable angina
* Left ventricular ejection fraction < 30%
* Valvular disease requiring interventional treatment
* Cardiac surgery within 3 months prior to enrolment
* Left atrial size > 55 mm as measured in the parasternal antero-posterior view
* Uncontrolled bleeding, diathesis, coagulopathy or pro-coagulant state
* Active systemic infection or sepsis
* Other co-morbid condition(s) that could limit the participant's ability to participate in the study or to comply with follow-up requirements, or impact the scientific integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Freedom from documented atrial tachyarrhythmia (every documented episode of atrial tachyarrhythmia lasting >/=30 seconds will be count as recurrence. | Month 12
  The primary endpoint of the current study is freedom from documented atrial tachyarrhythmia (>/=30 seconds) documented by ECG 4-12 months after PVI off antiarrhythmic drugs. Atrial tachyarrhythmias comprise AF as well as atrial tachycardia and atrial flutter.
  Holter-ECGs as well as 12-lead ECGs will be conducted. Every epsiode of documented atrial tachyarrhythmia (>/=30 seconds)outside the blanking period will count as "recurrence".

SECONDARY OUTCOMES:
Acute procedure success | Day 0
  Acute procedure success defined as the ability to confirm electrical isolation of the individual pulmonary vein with a circular mapping catheter (achieve catheter). Acute procedure success will be defined as pulmonary vein isolation of all target pulmonary veins.
  Pulmonary vein isolation will be detected by entrance block (absence of a pulmonary vein signal) on the circular mapping catheter.
Procedure duration | Intraoperative
  Procedure time (minutes)
Number of freeze-cycles to achive pulmonary vein isolation. | Day 0
  Number (n=x) of freeze-cycles to achive pulmonary vein isolation. For each PV the number of the freeze-cycles will be counted.
Radiation exposure of patient and operator | Day 0
  Radiation exposure of patient and operator (Gy/cm2)
Radiation exposure duration | Day 0
  Radiation exposure duration (minutes)
Periprocedural complications | Day 0
  Periprocedural complications (e.g. phrenic nerve injury, cardiac tamponade, groin injury etc.)
Duration of freeze-cycles to achive pulmonary vein isolation | Day 0
  Duration of freeze-cycles to achive pulmonary vein isolation (n=x)

CONTACTS AND LOCATIONS:
Locations (1):
- University Heart Center Luebeck, Electrophysiology, Lübeck, Germany